CLINICAL TRIAL: NCT04748926
Title: A Randomized, Open-label, Phase I Study to Assess the Effects of Food and Formulation on the Pharmacokinetics of a Single Dose of Rilzabrutinib (SAR444671 [Formerly PRN1008]) in Healthy Male and Female Participants
Brief Title: Food Effect and Relative Bioavailability Study of Rilzabrutinib in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Principia Biopharma, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PKM17098; U1111-1260-4526 (Other: UTN); PRN1008-25 (Other: Principia Biopharma)
Record Dates: First submitted 2021-02-03; First posted 2021-02-10 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): Participants will receive caplets after fast (treatment A) on Day 1 and caplets after meal (treatment B) on day 6, and then receive either oral formulation 1 tablets after fast (treatment C) or oral formulation 2 tablets after fast (treatment D) on day 11.
  Interventions: Drug: rilzabrutinib SAR444671
- Group 2 (Experimental): Participants will receive caplets after meal (treatment B) on Day 1 and caplets after fast (treatment A) on day 6, and then receive either oral formulation 1 tablets after fast (treatment C) or oral formulation 2 tablets after fast (treatment D) on day 11.
  Interventions: Drug: rilzabrutinib SAR444671

INTERVENTIONS:
Drug: rilzabrutinib SAR444671 — Pharmaceutical form: caplet Route of administration: oral
Drug: rilzabrutinib SAR444671 — Pharmaceutical form: Oral Formulation 1 tablets Route of administration: oral
Drug: rilzabrutinib SAR444671 — Pharmaceutical form: Oral Formulation 2 tablets Route of administration: oral

SUMMARY:
Primary Objective:

* To evaluate the impact of food on the pharmacokinetics (PK) of rilzabrutinib following single oral doses to healthy subjects.
* To evaluate the impact of formulation on the PK of rilzabrutinib following single oral doses to healthy subjects

Secondary Objective:

- To assess the safety and tolerability of single oral doses of rilzabrutinib administered under fasted and fed conditions

DETAILED DESCRIPTION:
The total study duration is approximately 43 days for each participant, including a screening period of 2 to 28 days, treatment period of 12 days, and follow-up of 3 days

ELIGIBILITY:
Inclusion criteria :

- Participants who are overtly healthy as determined by medical evaluation

* Body mass index (BMI) within the range ≥18 and ≤31 kg/m2 (inclusive) and a minimum body weight of 45 kg.
* Female participant is eligible to participate if she is not pregnant or breastfeeding
* Male participants are eligible to participate if they agree to refrain from donating sperm and use contraception/barrier or be abstinent from intercourse

Exclusion criteria:

* COVID-19 infection, positive test result for human immunodeficiency virus (HIV), hepatitis B virus or hepatitis C virus antibody
* Use of any prescription or over-the-counter (OTC) medication, herbal products, or dietary supplements within 7 days
* Participation in another clinical trial of a drug or device whereby the last investigational drug/device administration is within 30 days or 5 half-lives, whichever is longer, prior to the first dose of study drug.
* Clinically significant abnormal in vital signs. - Any specific situation during study implementation/course that may rise ethics considerations.

The above information is not intended to contain all considerations relevant to a subject's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-05-21 (Actual)

PRIMARY OUTCOMES:
Rilzabrutinib plasma PK parameters following administration of the reference formulation in the fed and fasted states: Cmax | From Day 1 to Day 7
  maximun plasma concentration
Rilzabrutinib plasma PK parameters following administration of the reference formulation in the fed and fasted states: Tmax | From Day 1 to Day 7
  time to maximum plasma concentration
Rilzabrutinib plasma PK parameters following administration of the reference formulation in the fed and fasted states: AUC0-last | From Day 1 to Day 7
  area under the plasma concentration-time curve from zero to the last measurable concentration
Rilzabrutinib plasma PK parameters following administration of the reference formulation in the fed and fasted states: AUC0-inf | From Day 1 to Day 7
  area under the plasma concentration-time curve from zero to infinity
Rilzabrutinib plasma PK parameters following administration of the reference formulation in the fed and fasted states: half-life | From Day 1 to Day 7
  terminal elimination phase half-life
Rilzabrutinib plasma PK parameters following administration of two test formulations in the fasted state: Cmax | From Day 11 to Day 12
  maximun plasma concentration
Rilzabrutinib plasma PK parameters following administration of two test formulations in the fasted state: Tmax | From Day 11 to Day 12
  time to maximum plasma concentration
Rilzabrutinib plasma PK parameters following administration of two test formulations in the fasted state: AUC0-last | From Day 11 to Day 12
  area under the plasma concentration-time curve from zero to the last measurable concentration
Rilzabrutinib plasma PK parameters following administration of two test formulations in the fasted state: AUC0-inf | From Day 11 to Day 12
  area under the plasma concentration-time curve from zero to infinity
Rilzabrutinib plasma PK parameters following administration of two test formulations in the fasted state: half-life | From Day 11 to Day 12
  terminal elimination phase half-life

SECONDARY OUTCOMES:
Treatment-emergent AE and treatment-emergent SAE | Until Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site, Adelaide, Australia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: PKM17098 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25326&tenant=MT_SNY_9011